CLINICAL TRIAL: NCT01054989
Title: Fat, Inflammation and Insulin Resistance (FIRE-Study)
Brief Title: Fat, Inflammation and Insulin Resistance
Acronym: FIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Principal Investigator, julia szendrödi, Julia Szendrödi, MD, PhD, German Diabetes Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FIRE-01
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Healthy Adults With Normal BMI
Keywords: Healthy adults; Insulin sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fat intravenously (Active Comparator): Intravenous application of fat
  Interventions: Biological: Fat/Inflammation effects
- Fat orally (Active Comparator): Oral fat load
  Interventions: Biological: Fat/Inflammation effects
- LPS intravenously (Active Comparator): Lipopolysaccharide (LPS; US Standard Reference endotoxin)
  Interventions: Biological: Fat/Inflammation effects
- Glycerol intravenously (Placebo Comparator): Intrevenous glycerol infusion
  Interventions: Biological: Fat/Inflammation effects

INTERVENTIONS:
Biological: Fat/Inflammation effects — Fat infusion (Intralipid) over 6 hours Fat orally (Soy bean oil) single dose LPS infusion for 10 minutes Glycerol infusion over 6 hours

SUMMARY:
The combination of impaired insulin sensitivity and insulin secretion is thought to be the basis of type 2 diabetes. Increased free fatty acids levels impair insulin action in muscle and liver, but also systemic inflammation processes play a role in the development of insulin resistance.

This study compares the effects of fat and inflammation on insulin sensitivity, systemic inflammation, energy metabolism, vascular system and neural function in healthy humans.

DETAILED DESCRIPTION:
A dysregulation of lipid metabolism with increased levels of free fatty acids (FFA) is known represent one key mechanism in the pathophysiology of insulin resistance, which is subsequently known to be the basis of the development of type 2 diabetes. But also inflammatory processes, also known as subclinical inflammation, have been shown to be independently associated with insulin resistance and diabetes development. The aim of this study is to analyse the causal relationship between FFA and inflammation in the induction of insulin resistance in healthy humans.

It is known that the parenteral application of lipids over 4-6 hours results in an increase of FFA and a subsequent induction of a transient insulin resistance in peripheral tissues. Whether oral fat intake has similar effect is still unknown. On the other hand the oral intake of a high fat meal acutely increases intestinal permeability and thereby the levels of bacterial lipopolysaccharide (LPS) in the bloodstream. LPS is known to be a potent stimulator of immune response on a subclinical level accompanied by elevated levels of immune mediators, which in turn impair the insulin receptor signalling pathway leading to insulin resistance. Thus, in this study the effects of fat, both by an oral or parenteral fat load, and by a short-term LPS-infusion simulating the postprandial systemic LPS peak compared to a control infusion (glycerol) on insulin resistance is analysed. Insulin resistance and hepatic glucose production is determined by an hyperinsulinemic euglycemic clamp including glucose tracers. To detect the effects on the immune system on different levels, we measure 1) circulating levels of immune mediators by ELISA and bead-based mulitiplex assays, 2) gene expression of leukocytes, 3) subfractions of circulating leukocytes by FACS and 4) the stimulatory capacity of isolated lymphocytes and monocytes in vitro. Moreover, the effects of fat or inflammation on the function of the autonomic nervous system and the vasculature are studied. A second focus is the impact of the interventions on signal transduction and mitochondrial function in muscle and as well as on the metabolism and inflammation in subcutaneous adipose tissue in muscle and fat biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Age 20-40
* BMI 20-25 mg/m2

Exclusion Criteria:

* Hyperlipidemia
* Smoking
* Pregnancy
* Acute infection
* Anaemia
* Taking drugs influencing lipid or glucose metabolism, the immune system or antihypertensive medication
* Malignancies
* Any chronic disease
* Autoimmune or immune compromising diseases including HIV/AIDS
* Allergies against study drugs
* Hepatitis
* Gall bladder diseases
* Renal failure
* Psychiatric diseases or addiction

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03-15 (Actual); Primary Completion 2011-09-15 (Actual); Study Completion 2012-10-15 (Actual)

PRIMARY OUTCOMES:
Effect of intervention on whole body insulin sensitivity | 6 hours

SECONDARY OUTCOMES:
Effect of intervention on systemic inflammation | 1-6 hours
Effect of intervention on cellular immune mechanisms | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Study Director — German Diabetes Center; Bettina Nowotny, MD, Principal Investigator — German Diabetes Center

REFERENCES:
- [Derived] Ziegler D, Strom A, Strassburger K, Nowotny B, Zahiragic L, Nowotny PJ, Carstensen-Kirberg M, Herder C, Szendroedi J, Roden M. Differential Patterns and Determinants of Cardiac Autonomic Nerve Dysfunction during Endotoxemia and Oral Fat Load in Humans. PLoS One. 2015 Apr 20;10(4):e0124242. doi: 10.1371/journal.pone.0124242. eCollection 2015. PMID 25893426
- [Derived] Nowotny B, Zahiragic L, Krog D, Nowotny PJ, Herder C, Carstensen M, Yoshimura T, Szendroedi J, Phielix E, Schadewaldt P, Schloot NC, Shulman GI, Roden M. Mechanisms underlying the onset of oral lipid-induced skeletal muscle insulin resistance in humans. Diabetes. 2013 Jul;62(7):2240-8. doi: 10.2337/db12-1179. Epub 2013 Mar 1. PMID 23454694